CLINICAL TRIAL: NCT00538681
Title: Randomized, Double-Blind, Placebo Controlled, Phase 2 Study of Pemetrexed and Cisplatin Plus Enzastaurin Versus Pemetrexed and Cisplatin Plus Placebo in Chemonaive Patients With Advanced, Unresectable, or Metastatic (Stage IIIB or IV) Nonsquamous Non-Small Cell Lung Cancer
Brief Title: Study for Participants With Advanced, Not Amenable to Surgery, or Metastatic Lung Cancer Comparing Treatment With Pemetrexed + Cisplatin + Enzastaurin Versus Pemetrexed + Cisplatin + Placebo
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to lack of efficacy demonstrated in relevant participant population in other clinical trials.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10722; H6Q-MC-S021 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-10-01; First posted 2007-10-03 (Estimated); Results first posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — enzastaurin; Pemetrexed; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enzastaurin + Pemetrexed + Cisplatin (Experimental)
  Interventions: Drug: enzastaurin; Drug: pemetrexed; Drug: cisplatin
- Placebo + Pemetrexed + Cisplatin (Placebo Comparator)
  Interventions: Drug: pemetrexed; Drug: cisplatin; Drug: placebo

INTERVENTIONS:
Drug: enzastaurin — 1125 milligrams (mg) loading dose then 500 mg, oral (po), daily (QD), until disease progression
  Other Names: LY317615
  Arms: Enzastaurin + Pemetrexed + Cisplatin
Drug: pemetrexed — 500 milligrams/square meter (mg/m²), intravenously (IV), every 21 days, for each 21-day cycle
  Other Names: LY231514; Alimta
Drug: cisplatin — 75 mg/m², IV, every 21 days, for each 21-day cycle
Drug: placebo — po, QD
  Arms: Placebo + Pemetrexed + Cisplatin

SUMMARY:
This study is intended for participants with advanced, not amenable to surgery, or metastatic lung cancer who have not received any prior chemotherapy. The study will be conducted in 2 parts:

* Part 1 is intended to evaluate safety of pemetrexed + cisplatin + enzastaurin combination chemotherapy
* Part 2 whose main objective is to compare the efficacy of pemetrexed + cisplatin + enzastaurin versus pemetrexed + cisplatin + placebo. Participants to be included in Part 2 are those with Nonsquamous Non-Small Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of advanced NSCLC not amenable to curative treatment. Participants enrolling in Part 2 of the study must have the above stated diagnosis of NSCLC that is also of nonsquamous histology.
* no prior systemic therapies [chemotherapy, et cetera (etc.)] or pleurodesis with chemotherapy for this disease
* prior radiotherapy is allowed but must be completed at least 2 weeks before study enrollment and participant must be recovered from the acute toxic effects
* have a good performance status
* participant must sign an informed consent document

Exclusion Criteria:

* participant had myocardial infarction occurring less than 6 months before inclusion, uncontrolled arrhythmia, symptomatic angina pectoris, or cardiac failure not controlled by medications
* participant is unable to swallow tablets
* participant is taking a certain medicine to control seizure activity, called "enzyme inducing antiepileptic drugs" and is not able to stop taking the medicine prior to enrolling in the study
* participant is unable to interrupt aspirin and/or other anti-inflammatory agents
* participant is unwilling or unable to take vitamin supplementation (folic acid and vitamin B12) or medications to prevent side effects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UCT/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven, Belgium
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gauting
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., GroBhansdorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Catania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trento
- Poland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Otwock
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest, Romania

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1- Cohort 1: Cycle 1: 500 milligrams (mg) enzastaurin orally (po) as loading dose on Day 1 and 125 mg orally twice daily (BID) on Days 2 to 28 of 28-day cycle then 500 milligrams per square meter (mg/m²) pemetrexed intravenous (IV) followed by 75 mg/m2 cisplatin IV on Day 8 of a 28-day cycle.
  Cycles 2 to 6: 125 mg enzastaurin po BID Days 1 to 21 of each 21-day cycle, then 500 mg/m² pemetrexed IV followed by 75 mg/m² cisplatin IV on Day 1 of each 21-day cycle.
- Part 1- Cohort 2: Cycle 1: 1125 mg enzastaurin po as loading dose on Day 1 of a 28-day cycle and 250 mg po BID on Days 2 to 28 of 28-day cycle, then 500 mg/m2 pemetrexed IV followed by 75 mg/m² cisplatin IV on Day 8 of a 28-day cycle.
  Cycles 2 to 6: 250 mg enzastaurin po BID Days 1 to 21 of each 21-day cycle, then 500 mg/m² pemetrexed IV followed by 75 mg/m² cisplatin IV on Day 1 of each 21-day cycle.
- Part 2- Enzastaurin: Cycle 1: 375 mg enzastaurin po 3 times on Day 1 as a loading dose and 250 mg po BID on Day 2 to 28 of a 28-day cycle, then 500 mg/m² IV followed by 75 mg/m² cisplatin IV on Day 8 of a 28-day cycle.
  Cycle 2 to 6: 250 mg enzastaurin po BID on Days 1 to 21 of each 21-day cycle, then 500 mg/m² pemetrexed IV followed by 75 mg/m² cisplatin IV on Day 1 of each 21-day cycle.
- Part 2- Placebo: Cycle 1: Placebo was administered po 3 times on Day 1 and BID on Days 2 to 28 of a 28-day cycle then 500 mg/m² pemetrexed followed by 75 mg/m² cisplatin administered IV on Day 8 of 28-day cycle.
  Cycle 2 to 6: Placebo was administered po BID on Days 1 to 21 of each 21-day cycle then 500 mg/m² pemetrexed followed by 75 mg/m² cisplatin administered IV on Day 1 of each 21-day cycle.
Period: Overall Study
Arm/Group | Part 1- Cohort 1 | Part 1- Cohort 2 | Part 2- Enzastaurin | Part 2- Placebo
Started | 9 | 4 | 11 | 11 (One (1) participant received pemetrexed and cisplatin only before the study was closed.)
Received ≥1 Dose of Any Study Drug | 9 | 4 | 11 | 11
Completed | 0 | 0 | 0 | 0
Not Completed | 9 | 4 | 11 | 11
Not completed — Progressive Disease | 7 | 0 | 1 | 0
Not completed — Sponsor Decision | 1 | 3 | 8 | 9
Not completed — Adverse Event | 1 | 1 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Investigator Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of any study drug.
Groups:
- Part 1- Cohort 1: Cycle 1: 500 mg enzastaurin orally (po) as loading dose on Day 1 and 125 mg orally twice daily (BID) on Days 2 to 28 of 28-day cycle then 500 milligrams per square meter (mg/m²) pemetrexed intravenous (IV) followed by 75 mg/m2 cisplatin IV on Day 8 of a 28-day cycle.
  Cycles 2 to 6: 125 mg enzastaurin po BID Days 1 to 21 of each 21-day cycle, then 500 mg/m² pemetrexed IV followed by 75 mg/m² cisplatin IV on Day 1 of each 21-day cycle.
- Other: 500 mg/m² pemetrexed and 75 mg/m² cisplatin administered intravenously
- Total: Total of all reporting groups
Arm/Group | Part 1- Cohort 1 | Part 1- Cohort 2 | Part 2- Enzastaurin | Part 2- Placebo | Other | Total
Number analyzed (Participants) | 9 | 4 | 11 | 10 | 1 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (9.32) | 61.2 (6.85) | 58.6 (9.62) | 59.5 (9.39) | 49.1 (NA) — Only 1 participant in the group | 58.8 (8.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 6 | 6 | 1 | 16
  Male | 8 | 2 | 5 | 4 | 0 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 9 | 4 | 11 | 10 | 1 | 35
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 4 | 1 | 1 | 4 | 0 | 10
  Poland | 0 | 0 | 4 | 4 | 1 | 9
  Germany | 5 | 3 | 6 | 2 | 0 | 16
Type of Carcinoma [Count of Participants; unit: Participants]
  Adenocarcinoma: Lung | 7 | 3 | 1 | 4 | 0 | 15
  Carcinoma Large Cell: Lung | 1 | 0 | 3 | 2 | 0 | 6
  Squamous Cell Carcinoma: Lung | 1 | 1 | 0 | 0 | 0 | 2
  Carcinoma Non-Small Cell: Lung | 0 | 0 | 2 | 1 | 0 | 3
  Adenocarcinoma, Bronchioalveolar | 0 | 0 | 5 | 3 | 1 | 9
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG classifies participants according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  Participants
    0-Fully Active | 1 | 1 | 4 | 3 | 0 | 9
    1-Ambulatory, work of a light or sedentary nature | 8 | 3 | 7 | 7 | 1 | 26

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Evaluate Safety [Toxicity, Serious Adverse Events (SAEs) and Reasons for Participant's Discontinuation]
Description: Presented are data that evaluates safety based on toxicity using Common Terminology Criteria for Adverse Events (CTCAE v3.0), SAEs, and discontinuations due to SAEs or other non-serious adverse events (AE's) of study participants. A summary of SAEs and other non-serious AEs regardless of causality is located in the Reported Adverse Event module.
Time Frame: Cycle 1 (28-day cycle), Cycles 2, 3, 4, 5, and 6 (21-day cycles) and 30-day follow up
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Cohort 1 | Part 1- Cohort 2
Number analyzed (Participants) | 9 | 4
Participants
  SAEs | 5 | 0
  AEs | 9 | 4
  Discontinued due to AE | 1 | 1

2. Primary Outcome: Part 2: Compare Progression-Free Survival (PFS) Between the 2 Treatment Arms Through the Assessment of Tumor Response
Description: PFS was defined as the time from date of first dose to the first observation of disease progression or death due to any cause. For participants not known to have died as of the data cut-off date and who did not have objective progressive disease (PD), PFS was censored at the date of the last objective progression-free assessment. For participants who received subsequent anticancer therapy (after discontinuation from the study treatment) prior to objective disease progression or death, PFS was censored at the date of last objective progression-free assessment prior to the initiation of post discontinuation anticancer therapy. PFS was calculated and analyzed based on an alternative definition of censoring; for each participant who is not known to have died or who have had objective disease progression as of the data cut-off date, PFS was censored at the date of last prior contact. Zero participants were analyzed in this outcome as study was terminated early.
Time Frame: Baseline to measured PD up to 5 months
Population: No participant completed a full cycle of therapy and data were not collected for this Outcome Measure.
Groups:
- Part 2- Enzastaurin: Cycle 1: 375 milligrams (mg) enzastaurin orally (po) 3 times on Day 1 as a loading dose and 250 mg po twice daily (BID) on Day 2 to 28 of a 28-day cycle, then 500 milligrams per square meter (mg/m²) intravenous (IV) followed by 75 mg/m² cisplatin IV on Day 8 of a 28-day cycle.
  Cycle 2 to 6: 250 mg enzastaurin po BID on Days 1 to 21 of each 21-day cycle, then 500 mg/m² pemetrexed IV followed by 75 mg/m² cisplatin IV on Day 1 of each 21-day cycle.
Arm/Group | Part 2- Enzastaurin | Part 2- Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Part 2: To Evaluate the Safety and Toxicity Profile of Study Treatments
Description: The safety and toxicity profile for Part 2 was defined as serious adverse events (SAEs) and other non-serious adverse events (AEs). A summary of SAEs and other non-serious AEs regardless of causality is located in the Reported Adverse Event module.
Time Frame: Cycle 1 (28-day cycle), Cycles 2, 3, 4, 5, and 6 (21-day cycles) and 30-day follow-up
Population: All randomized participants who received at least 1 dose enzastaurin or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2- Enzastaurin | Part 2- Placebo
Number analyzed (Participants) | 11 | 10
Participants
  SAEs | 2 | 4
  AEs | 8 | 8

4. Secondary Outcome: Part 2: Number of Participants With a Complete Response (CR) or Partial Response (PR) (Response Rate)
Description: Response rate was defined using Response Evaluation Criteria in Solid Tumors (RECIST v1.0) criteria. Complete Response (CR) was defined as the disappearance of all target lesions. Partial Response (PR) was defined as having at least a 30% decrease in sum of longest diameter (LD) of target lesions. Best response was confirmed by a second assessment in ≥28 days. Response rate was defined as the number of participants with best response of CR or PR divided by the total number of treated participants. Zero participants were analyzed in this outcome as study was terminated early.
Time Frame: Baseline to measured progressive disease (PD) up to 5 months
Population: No participant completed a full cycle of therapy and data were not collected for this Outcome Measure.
Arm/Group | Part 2- Enzastaurin | Part 2- Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Part 2: Overall Survival (OS)
Description: OS time was defined as the time from the date of study enrollment to the date of death from any cause. For participants not known to have died as of the data cut-off date, OS was censored at the last contact date (last contact for participants in post discontinuation was equal to the last known alive date in mortality status). Zero participants were analyzed in this outcome as study was terminated early.
Time Frame: Baseline to date of death from any cause up to 5 months
Population: No participant completed a full cycle of therapy and data were not collected for this Outcome Measure.
Arm/Group | Part 2- Enzastaurin | Part 2- Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Part 2: Duration of Disease Control (DDC) and Response
Description: DDC and response defined as time from complete response (CR), partial response (PR) or stable disease (SD) to first date of objectively determined progressive disease (PD) or death from any cause using RECIST (v1.0) criteria. CR defined as disappearance of all target lesions. PR defined as having ≥30% decrease in sum of longest diameter (LD) of target lesions. PD defined as having ≥20% increase in the sum of the LD of target lesions. SD defined as small changes not meeting above criteria. Participants not known to have died as of data cut-off date, had no objective PD or were lost to follow-up, DCC was censored at date of last objective progression-free assessment (OPFA). Participants who received subsequent anticancer therapy (after discontinuation from study treatment) prior to objective PD or death were censored at date of last OPFA prior to initiation of post discontinuation anticancer therapy. Zero participants were analyzed in this outcome as study was terminated early.
Time Frame: Baseline to measured PD up to 5 months
Population: No participant completed a full cycle of therapy and data were not collected for this Outcome Measure.
Arm/Group | Part 2- Enzastaurin | Part 2- Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Part 2: Time to Worsening of Symptoms (TWS)
Description: TWS was measured from the date of study enrollment to the first date of a worsening in any of the 6 Lung Cancer Symptom Scale (LCSS) symptoms (appetite, cough, fatigue, shortness of breath, hemoptysis and pain). Participants marked each symptom on a visual analog scale (VAS) that ranged from 0 millimeter (mm) (as good as it can be/none) to 100 mm (as bad/much as it could be). TWS was also measured individually for each of the 6 symptoms independently and were also measured from the date of enrollment to the first date of worsening in pain. For both measurements, worsening was defined as a 15-mm increase from baseline in the participant-reported score for any symptom. Participants who are not known to have had a worsening TWS were censored at the date of the participant's last LCSS assessment. Zero participants were analyzed in this outcome as study was terminated early.
Time Frame: Cycle 1 (28-day cycle), Cycles 2, 3, 4, 5, and 6 (21-day cycles) and 30-day follow-up
Population: No participant completed a full cycle of therapy and data were not collected for this Outcome Measure.
Arm/Group | Part 2- Enzastaurin | Part 2- Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Part 2: To Assess Biomarkers of the Disease State and Their Correlation to Clinical Outcome
Description: Presented are data that evaluates of biomarkers relevant to the study drug and the disease state of the participant's clinical outcome. Zero participants were analyzed in this outcome as study was terminated early.
Time Frame: Baseline, Cycle 1 (28-day cycle), Cycles 2, 3, 4, 5, and 6 (21-day cycles) and end of study up to 5 months
Population: No participant completed a full cycle of therapy and data were not collected for this Outcome Measure.
Arm/Group | Part 2- Enzastaurin | Part 2- Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Study-specific clinical outcomes due to progressive disease (PD) were not considered to be a serious adverse event (SAE) unless the investigator deemed it related to the use of the study drug.
Groups:
- Part 1- Cohort 1: Cycle 1: 500 mg Enzastaurin orally as loading dose on Day 1 of a 28-day cycle and 125 mg orally twice daily, plus 500 mg/m2 pemetrexed intravenous (IV) and 75 mg/m2 cisplatin IV on Day 8 of a 28-day cycle.
  Cycles 2-6: 125 mg Enzastaurin orally twice daily, with 500 mg/m2 pemetrexed IV and 75 mg/m2 cisplatin IV on Day 1 of each 21-day cycle.
- Part 1- Cohort 2: Cycle 1: 1125 mg Enzastaurin orally as loading dose on Day 1 of a 28-day cycle and 250 mg orally twice daily starting on Day 2, plus 500 mg/m2 pemetrexed IV and 75 mg/m2 cisplatin IV on Day 8 of a 28-day cycle.
  Cycles 2-6: 250 mg Enzastaurin orally twice daily, with 500 mg/m2 pemetrexed IV and 75 mg/m2 cisplatin IV on Day 1 of each 21-day cycle.
- Part 2- Enzastaurin: Cycle 1: 375 mg Enzastaurin orally 3 times on Day 1 of a 28-day cycle and 250 mg orally twice daily starting on Day 2, plus 500 mg/m² pemetrexed intravenously (IV) and 75 mg/m² cisplatin IV on Day 8 of a 28-day cycle.
  Cycle 2-6: 250 mg Enzastaurin orally twice daily on Days 1 to 21 (21-day cycles) with 500 mg/m² pemetrexed IV and 75 mg/m² cisplatin IV on day 1 of each 21-day cycle.
- Part 2- Placebo: Cycle 1: Placebo was administered orally 3 times on Day 1 and 2 times a day on Days 2-28 (28-day cycle) plus 500 mg/m² pemetrexed IV and 75 mg/m² cisplatin IV on Day 8 of cycle (28-day cycle).
  Cycle 2-6: Placebo was administered orally 2 time a day on Days 1 to 21 (21-day cycles) plus 500 mg/m² pemetrexed IV and 75 mg/m² cisplatin IV on Day 1 of each 21-day cycle.
- Part 2- Pemetrexed + Cisplatin: Participant was not randomized to Arm A or Arm B but received 500 mg/m² pemetrexed and 75 mg/m² cisplatin administered intravenously but not randomized
Arm/Group | Part 1- Cohort 1 | Part 1- Cohort 2 | Part 2- Enzastaurin | Part 2- Placebo | Part 2- Pemetrexed + Cisplatin
Serious Adverse Events (participants affected / at risk) | 5/9 | 0/4 | 2/11 | 4/10 | 0/1
Other Adverse Events (participants affected / at risk) | 9/9 | 4/4 | 8/11 | 8/10 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1- Cohort 1 (N=9) | Part 1- Cohort 2 (N=4) | Part 2- Enzastaurin (N=11) | Part 2- Placebo (N=10) | Part 2- Pemetrexed + Cisplatin (N=1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1- Cohort 1 (N=9) | Part 1- Cohort 2 (N=4) | Part 2- Enzastaurin (N=11) | Part 2- Placebo (N=10) | Part 2- Pemetrexed + Cisplatin (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual disturbance (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (5) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (8) | 3 (11) | 3 (5) | 5 (7) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (7) | 2 (4) | 3 (4) | 2 (3) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 7 (7) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 6 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neutrophil count (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Urine colour abnormal (Investigations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This trial was terminated due to lack of efficacy demonstrated in relevant participant population in other clinical trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days